CLINICAL TRIAL: NCT06905210
Title: Phase III Superiority, Randomized, Double-blind, Placebo-controlled, Adaptive, Multicenter Study to Compare the Efficacy and Safety of a New Concentration of an Antiandrogenic Progestogen Combined With a Reduced-dose Estrogen for the Treatment of Moderate Acne Vulgaris
Brief Title: Study of New Antiandrogenic Progestogen + Low-dose Estrogen for Moderate Acne Vulgaris
Acronym: PANDORA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EF190
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Acne Vulgaris; Acne Vulgaris on the Face
Keywords: Acne treatment; fixed-dose combination; moderate acne; randomized controlled trial; women's dermatology; adaptive clinical study; efficacy & safety evaluation; hormonal acne research; Moderate acne vulgaris; Phase III; Randomized; Double-blind; Placebo-controlled; Adaptive design; Multicenter; Superiority trial
MeSH Terms: conditions — Acne Vulgaris | interventions — Drugs, Investigational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Drug: Experimental drug
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo of the experimental drug

INTERVENTIONS:
Drug: Placebo of the experimental drug — Subjects randomized to this group will receive one (01) placebo of the experimental drug everyday for 28 weeks.
  Arms: Placebo Group
Drug: Experimental drug — Subjects randomized to this group will receive one (01) experimental drug everyday for 28 weeks.
  Arms: Experimental Group

SUMMARY:
This Phase III randomized, double-blind, placebo-controlled, adaptive, multicenter study evaluates the efficacy and safety of a new concentration of the fixed-dose combination EF190 in women with moderate acne vulgaris over six 28-day treatment cycles. Eligible participants will be randomized (2:1) to receive either the experimental drug or placebo alongside standard skincare. The study includes five in-person visits (screening, randomization, and three follow-ups) and three phone contacts (cycles 2, 4, and 5) to monitor adherence, adverse events, and contraceptive use. A subgroup will undergo additional exploratory assessments, including acne questionnaires, ovarian activity tests, photographic documentation, and specialized lab/ultrasound exams.

DETAILED DESCRIPTION:
This is a Phase III, randomized, double-blind, placebo-controlled, adaptive, multicenter superiority study to evaluate the efficacy and safety of a new concentration of the fixed-dose combination EF190 in women with moderate acne vulgaris after six treatment cycles. Eligible participants will be randomized into a controlled, double-blind treatment period, receiving either the experimental drug or placebo, along with standard skin care, for six 28-day cycles.

Throughout the study, each participant must attend at least five (05) in-person clinic visits at the research center. At the screening visit (VS/V1), the participant will sign the Informed Consent Form (ICF) and the Assent Form (AF), undergo eligibility assessment, and have blood drawn. At the randomization visit (VR/V2), eligibility will be confirmed, baseline acne data (lesions and score) will be recorded, randomization (2:1 for treatment/placebo) will occur, and the study medication will be dispensed. The first dose (Day 1) will be administered on the 28th day post-menstruation. Subsequent visits (V3-V5/VF) will take place on day 15 (±3) of each cycle. The final visit (V5/VF) will assess the study's primary endpoint.

In addition to in-person visits, participants will have three (3) phone contacts, scheduled between clinic visits during cycles 2, 4, and 5. These calls aim to reinforce treatment adherence, collect information on adverse events and concomitant medications, assess discontinuation criteria, and remind participants about the use of study-permitted contraceptive methods.

Furthermore, a subgroup of participants will be selected for exploratory evaluations. These participants will complete acne control questionnaires, undergo ovarian activity assessments, have photographic documentation for acne evaluation, and receive specified laboratory and ultrasound tests as per the protocol and ICF/AF.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to confirm voluntary participation and agree to all trial procedures by signing the Informed Consent Form (ICF) and Informed Assent Form (ITA), if applicable, prior to any procedure provided for in the protocol. Note: The adult participant or the participant's guardian when the participant is a legal minor (adolescent) must sign the ICF after understanding and agreeing to all trial procedures. The adolescent participant must provide assent by signing the ITA based on local regulations and/or guidelines prior to the start of any study procedures.
2. Female sex.
3. Age between 14 and 45 years (inclusive).
4. At least one year after menarche.
5. At least one menstrual period during the last 03 months.
6. Absence of known contraindications for the use of combined oral contraceptives. 7. Diagnosis of moderate acne vulgaris on the face for at least six months, characterized by the presence of:

Note: Information regarding the duration of the disease can be obtained from the clinical history reported by the participant or from a brief medical report of the participant's history, if she is referred from another service.

1. At least 15 inflammatory lesions (papules or pustules);
2. At least 10 non-inflammatory lesions (comedones); and
3. Up to 03 small inactive nodules. Note: Nodules are lesions between 10 and 30 mm, more palpable than visible.

   8. Classification ≥ 3 on the 6-point scale of the Investigator's Static Global Assessment (ISGA).

   9. When the participant did not obtain adequate results with topical treatment, failure or impossibility of systemic treatment with antibiotics (contraindications or intolerance) and the patient has an indication for the use of antiandrogens and/or isotretinoin.

   10. Agreement not to use other topical and/or systemic treatments for acne during the study.

Exclusion Criteria:

1. Confirmed or suspected pregnancy. 2. History of childbirth, abortion or lactation in the last 3 months. 3. Participants who do not agree to use non-hormonal contraceptive methods permitted during the study, unless they are surgically sterile or who expressly declare themselves to be free from risk of pregnancy because they do not engage in sexual practices or engage in them in a non-reproductive manner.

4. Current or previous treatment with agents described below with a washout period shorter than that provided for each:

1. At least 6 months for systemic isotretinoin and/or injectable contraceptive (such as Depo Provera);
2. At least 3 months for implantable contraceptives (such as Implanon) or Levonorgestrel-Releasing Intrauterine System (such as Mirena and Kyleena);
3. At least 2 months for oral contraceptives or other systemic anti-acne agents not mentioned (such as systemic antibiotics);
4. At least 4 weeks for topical retinoids;
5. At least 2 weeks for other topical anti-acne agents (such as topical antibiotics or benzoyl peroxide); 5. Personal history or first-degree family history of vascular disease including previous arterial thromboembolic disease (myocardial infarction or stroke), venous thromboembolic disease (peripheral venous thrombosis or pulmonary embolism) or any condition that increases the risk for any of the previous conditions.

   6. Known personal history of thrombophilia. 7. Current smoking. 8. Any disease or condition that compromises the function of body systems that would result in altered absorption, excessive accumulation, impaired metabolism or altered excretion of the study medication, including malabsorptive conditions (such as previous bariatric surgery).

   9. Any condition that worsens under hormonal treatment or that interferes with the conduct of the study or interpretation of the results, such as gestational herpes or idiopathic jaundice during previous pregnancy, otosclerosis, Sydeham's chorea, porphyria, bile flow disorders (presence or history of cholestasis, gallstones, systemic lupus erythematosus).

   10. Other comorbidities (history or current diagnosis) such as chronic inflammatory bowel disease (Crohn's disease or ulcerative colitis), hemolytic uremic syndrome, headache with focal neurological symptoms, epilepsy, asthma with chronic use of oral corticosteroids, multiple sclerosis, Chorea minor, tetany, endometriosis, mastopathy, current premenstrual dysphoric disorder, sickle cell anemia, pancreatitis, vascular complications of diabetes, major depressive disorder or other conditions that, in the investigator's assessment, may compromise the participant's safety.

   11. Hypersensitivity to any of the components of the experimental drug or placebo.

   12. Presence of moderate to severe atopy, acne comedonica or acne conglobata, induced acne or acne with multiple large nodules, cysts, fistular comedones or fistular duct abscess or other dermatological conditions that, in the investigator's assessment, may compromise the evaluation of efficacy.

   13. Use of comedogenic creams or sunscreens, other preparations with sex hormones or any other anti-acne therapy (such as phototherapy, oleic acids, chemical peeling, mechanical extraction of comedones).

   14. Preparations with acnegenic effects, such as iodinated or brominated drugs, tuberculostatics, lithium, vitamins B1 (> 1.5 mg/day), B6 (> 2 mg/day) or B12 (> 6 g/day), corticosteroids, adrenocorticotropic hormone (ACHT), anabolic steroids, quinine, disulfiram, methoxypsoralen, phenobarbital, phenytoin, trimethadione, thyroid depressants, certain oily cosmetics.

   15. History of drug abuse. 16. History of neoplasia in the last 5 years, except non-melanoma skin cancer, or any history of sex hormone-dependent neoplasia or current suspicion of neoplasia, including meningioma.

   17. Use of other medications that interfere with hepatic metabolism via cytochrome P450, such as carbamazepine, phenytoin, primidone, oxcarbazepine, topiramate, rifampicin, ritonavir and products containing St. John's wort.

   18. Use of direct-acting antiviral medications containing ombitasvir, paritaprevir or dasabuvir and combinations of these medications.

   19. Undiagnosed vaginal bleeding. 20. Change in clinical breast examination or other clinically significant finding on gynecological examination that could, in the opinion of the investigator, be worsened by oral contraceptives. 21. Absence of proof of a Pap smear (oncotic cytology) without changes suspicious of malignancy in the last 12 months. Note: If the participant does not have a previous exam within the accepted interval and agrees, the exam may be performed at the Selection Visit (VS/V1).

   22. Absence of proof of a bilateral mammogram without changes suspicious of malignancy in the last 12 months, only for participants aged ≥ 40 years. Note: Mammograms with suspicious of malignancy are considered 23. Obesity (BMI > 30 kg/m²). 24. Uncontrolled arterial hypertension (Systolic Blood Pressure [SBP] ≥140 mmHg or Diastolic Blood Pressure [DBP] ≥ 90 mmHg).

   25. Participant who has participated in clinical trial protocols in the last 12 (twelve) months, unless the investigator believes that there may be direct benefit to the participant.

   26. Participant who, in the opinion of the investigator, presents other clinical or laboratory conditions or alterations that make him/her unfit to participate in the study

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 526 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the inflammatory lesion count at cycle 6. | 28 weeks
  Inflammatory lesion refears to open and closed comedones, papules, pustules, and nodules
Change from Baseline in the percentage of participants with scores 0 or 1 in the Static Investigator Global Assessment (ISGA) at cycle 6. | 28 weeks
  0 corresponds to "normal, clear skin with no evidence of acne vulgaris.";
  1 corresponds to "skin is almost clear: few non-inflammatory lesions present, with rare non-inflamed papules (papules must be resolving and may be hyperpigmented, though not pink-red). No nodular lesions are present."; 5 indicates "numerous highly inflammatory lesions predominate, with a variable number of comedones, many papules and pustules, or nodular lesions."

SECONDARY OUTCOMES:
Change from Baseline in the inflammatory lesion count at cycle 3. | 14 weeks
  Inflammatory lesion refears to open and closed comedones, papules, pustules, and nodules
Change from Baseline in the percentage of participants with scores 0 or 1 in the Static Investigator Global Assessment (ISGA) at cycle 3. | 14 weeks
  0 corresponds to "normal, clear skin with no evidence of acne vulgaris.";
  1 corresponds to "skin is almost clear: few non-inflammatory lesions present, with rare non-inflamed papules (papules must be resolving and may be hyperpigmented, though not pink-red). No nodular lesions are present."; 5 indicates "numerous highly inflammatory lesions predominate, with a variable number of comedones, many papules and pustules, or nodular lesions."
Absolute change from Baseline in the Acne-Specific Quality of Life Questionnaire (Acne-QoL) at cycle 3 and cycle 6. | 14 and 28 weeks
  The questionnaire has four (4) domains: Self perception (score range, 0 - 30), Role-Social (0 - 24), Role-emotional (0 - 30), and Acne Symptons (0 - 30). Overall, tem sum for all domains scores range from 0 to 114.
  Each domain scores responses are numbered starting with '0' in ascending order (ie. extremely=0, very much=1, quite a bit=2, a good bit=3, somewhat=4, a little bit=5, not at all=6). Higher scores for each domain in Acne-Specific Quality of Life Questionnaire (Acne-QoL) reflect increased health related quality of life, ie. less negative self perception, social, emotional and symptomatic effects associated with acne.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratórios S.A, Itapevi, São Paulo, Brazil